CLINICAL TRIAL: NCT04962555
Title: Clinical Related Study on Surgical Treatment of Knee Joint Meniscus Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-2015159
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Meniscus Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Meniscus Suture: The patient underwent meniscus suture surgery
  Interventions: Procedure: Meniscus Suture
- Partial meniscus resection: The patient underwent partial meniscus resection
  Interventions: Procedure: Partial meniscus resection
- Subtotal meniscus resection: The patient underwent Subtotal meniscus resection
  Interventions: Procedure: Subtotal meniscus resection
- Complete meniscectomy: The patient underwent complete meniscectomy
  Interventions: Procedure: Complete meniscectomy

INTERVENTIONS:
Procedure: Meniscus Suture — Patients with knee joint meniscus injury undergoing meniscus suture
  Groups: Meniscus Suture
Procedure: Partial meniscus resection — Patients with knee joint meniscus injury undergoing partial meniscus resection
  Groups: Partial meniscus resection
Procedure: Subtotal meniscus resection — Patients with knee joint meniscus injury undergoing subtotal meniscus resection
  Groups: Subtotal meniscus resection
Procedure: Complete meniscectomy — Patients with knee joint meniscus injury undergoing complete meniscectomy
  Groups: Complete meniscectomy

SUMMARY:
Through the analysis of the data of 8094 patients with knee meniscus injury before December 31, 2008 and more patients with partial meniscus resection, subtotal resection and total resection, we can understand the gender difference and ratio of medial and lateral meniscus injuries. Differences, differences in locations, differences in tearing methods, differences in surgical methods, and the course of the disease affect the meniscus injury and surgical methods, and further affect the patient's knee degeneration imaging, accompanying cartilage injury, knee osteoarthritis, Partial resection, subtotal resection and meniscus regeneration after total resection, imaging and secondary arthroscopic exploration (Second-Look) were studied.

DETAILED DESCRIPTION:
Through the data of 8094 patients with knee meniscus injury who underwent surgery at the Institute of Sports Medicine of the Third Hospital of Beijing Medical University before December 31, 2008, and the patients who underwent meniscus suture, partial resection, subtotal resection, and total resection. Analyze and understand the influence of gender difference, ratio difference, position difference, tearing method difference, surgical method difference and disease course on the meniscus injury situation and operation method of the internal and lateral meniscus injury. Observation and research will also be conducted on reports of knee cartilage injury, knee osteoarthritis, and meniscus regeneration after partial meniscus resection, subtotal resection and total resection.

ELIGIBILITY:
Inclusion Criteria:

Before December 31, 2008, patients who underwent surgery for meniscus injury in this institute and patients who underwent meniscus suture, partial resection, subtotal resection, and total resection.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 8778 patients with meniscus injury who underwent surgery at the Institute of Sports Medicine of the Third Hospital of Peking University before December 31, 2008 and patients who underwent meniscus suture, partial resection, subtotal resection, or total resection afterwards
Sampling Method: Probability Sample
Enrollment: 8778 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Meniscus injury site | During operation
  Observe the meniscus injury site during the operation, which is divided into: medial and lateral anterior horn, medial and lateral body, medial and lateral posterior horn, medial and lateral disc.
Types of Meniscus Injury | During operation
  The types of meniscus injuries were observed during the operation, which were divided into longitudinal fissure, oblique fissure, spallation, radial fissure, and barrel shank tear.
Meniscus surgery method | During operation
  Meniscus surgery methods include: partial resection, subtotal resection, total resection, and suture.
Cartilage damage | During operation
  The cartilage damage is evaluated as yes or no, where the cartilage surface is smooth and complete is defined as no, and the rest is defined as yes.
Cartilage damage | 7 years after surgery
  Second-look after operation to observe whether the cartilage is damaged. The cartilage damage is evaluated as yes or no, where the cartilage surface is smooth and complete is defined as no, and the rest is defined as yes.
Meniscus regeneration | 7 years after surgery
  Second-look after operation to observe whether the meniscus is regenerating. The Meniscus regeneration is evaluated as yes or no, in which the meniscus shape is complete and no tear is defined as yes, and other conditions are defined as no.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Prof., Study Chair — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China